CLINICAL TRIAL: NCT02370693
Title: Comparing and Combining Bortezomib and Mycophenolate in SSc Pulmonary Fibrosis Grant Number: R34HL122558
Brief Title: Comparing and Combining Bortezomib and Mycophenolate in SSc Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Manu Jain, Professor in Medicine-Pulmonary and Pediatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R34; 1R34HL122558-01A1 (NIH)
Record Dates: First submitted 2015-02-11; First posted 2015-02-25 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Lung Diseases, Interstitial; Systemic Sclerosis; Scleroderma
Keywords: mycophenolate; lung scarring
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Bortezomib; Saline Solution; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bortezomib plus mycophenolate mofetil (Active Comparator): Bortezomib 1.3 mg/m² subcutaneously (or IV push if unable to tolerate subcutaneous injection) once per week for the first two weeks per month and mycophenolate mofetil 1.5 g orally twice daily for 24 weeks
  Interventions: Drug: Bortezomib; Drug: Mycophenolate mofetil
- Placebo plus mycophenolate mofetil (Placebo Comparator): Placebo (normal saline) 1.3 mg/m² subcutaneously (or IV push if unable to tolerate subcutaneous injection) once per week for the first two weeks per month and mycophenolate mofetil 1.5 g orally twice daily for 24 weeks
  Interventions: Drug: Placebo; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.3 mg/m² subcutaneously (or IV push if unable to tolerate subcutaneous injection) once per week for the first two weeks per month for 24 weeks
  Other Names: Velcade
  Arms: bortezomib plus mycophenolate mofetil
Drug: Placebo — Placebo (normal saline) 1.3 mg/m² subcutaneously (or IV push if unable to tolerate subcutaneous injection) once per week for the first two weeks per month for 24 weeks
  Other Names: normal saline
  Arms: Placebo plus mycophenolate mofetil
Drug: Mycophenolate mofetil — Mycophenolate mofetil 1.5 g twice a day orally for 24 weeks
  Other Names: CellCept

SUMMARY:
The purpose of this study is to look at whether bortezomib, mycophenolate or the combination of both is better to treat scarring of the lung caused by Systemic Sclerosis.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a chronic multisystem autoimmune connective tissue disease for which the etiology remains unknown. The prevalence for SSc is between 19-75 cases per 100,000 and it is more frequent in women, with a peak occurrence in the 4th or 5th decade of life. Morbidity and Mortality in SSc are substantial and pulmonary complications are now the leading cause of death among patients with SSc.

Bortezomib is an FDA approved therapy for the treatment of multiple myeloma and other malignancies. The investigators have data that bortezomib inhibits transforming growth factor (TGF) - signaling in vitro and promotes normal repair and prevents against lung fibrosis in the TGF-mediated intratracheal bleomycin mouse model as well as in a mouse model for skin fibrosis. This is consistent with other data in the literature that proteasomal inhibition can prevent the development of fibrosis. Further there are multiple reports on the efficacy of bortezomib in ameliorating chronic graft-versus-host disease in patients after allogeneic hematopoietic stem cell transplant for multiple myeloma. Bortezomib was also well tolerated in the large clinical trials of multiple myeloma patients with neuropathy and thrombocytopenia the primary adverse events. No pulmonary toxicities were reported in these studies.

Mycophenolate mofetil (CellCept or Myfortic) belongs to a class of medications known as immunosuppressives. This medication was used originally in the management of patients with organ transplants, but is now recommended in the treatment of some autoimmune diseases such as SSc.

Mycophenolate mofetil targets an enzyme in the body called inosine monophosphate dehydrogenase that is important for the formation of deoxyribonucleic acid (DNA) in cells. By interfering with DNA, the medication impairs function of immune system cells that become overactive in autoimmune diseases. Mycophenolate mofetil is currently approved in the treatment of patients with SSc.

This study is being conducted to establish the safety and tolerability of bortezomib in SSc patients at high risk for pulmonary disease progression. In addition, the study will examine the effect of bortezomib on the rate of forced vital capacity (FVC) decline (a physiologic parameter closely associated with disease outcome) and other clinical parameters. In addition the investigators will also measure the effect of bortezomib on biomarkers associated with fibroblast activation. If successful, the study will provide the rationale for a multi-center placebo controlled trial to test the efficacy of bortezomib in SSc patients at high risk for progressive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Meet established criteria for diffuse or limited systemic sclerosis (SSc) and evidence of pulmonary at high risk of progression with or without progressive skin disease.
* Definition includes subjects who meet the American College of Rheumatology criteria for scleroderma
* High Risk of disease progression (see rationale) will be defined as follows
* If first non-Raynaud's manifestation of SSc < 36 months, then if any of the following are true: FVC <70% predicted or high-resolution computed tomography (HRCT) maximum fibrosis score >3 or FVC < 85% and modified Rodnan skin score (mRSS) increase > 5 over 6 months Regardless of disease duration
* Fall in FVC > 10% over the preceding 12 months or less in the absence of prior therapy or another identified causative process as assessed by the primary scleroderma physician
* Fall in FVC > 10% over 6 months on at least 12 months of prior therapy
* Age > 18 years
* Ability to give informed consent.
* Willingness to discontinue present therapy for the duration of the study
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* No evidence of acute infection
* Absolute neutrophil count >1000
* Platelets >75,000
* Stable mycophenolate mofetil dose for 16 weeks

Exclusion Criteria:

* Inability to give informed consent or comply with protocol procedures
* FVC < 40% or diffusing capacity of carbon monoxide (DLCO) <30% predicted
* Patient has a platelet count of less than 50,000 within 14 days before enrollment.
* Patient has an absolute neutrophil count of less 1000 within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of < 20 ml/minute within 14 days before enrollment.
* Patient has Grade 2 peripheral neuropathy by history within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum -human chorionic gonadotropin (- hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs within 4 weeks before enrollment
* Serious medical co-morbidity which in the opinion of the investigator makes participation in the study too high risk
* Psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03; Primary Completion 2019-12-16 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manu Jain, MD, MSc, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects were enrolled (signed consent form) but did not continue through the screening process far enough to reach randomization.
Period: Overall Study
Arm/Group | Bortezomib Plus Mycophenolate Mofetil | Placebo Plus Mycophenolate Mofetil
Started | 3 | 4
Completed | 2 | 3
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: 2 subjects were enrolled (signed consent form) but did not continue through the screening process far enough to reach randomization.
Groups:
- Enrolled But Not Randomized: Subjects who were enrolled (signed consent form) but did not continue through the screening process far enough to reach randomization.
- Total: Total of all reporting groups
Arm/Group | Bortezomib Plus Mycophenolate Mofetil | Placebo Plus Mycophenolate Mofetil | Enrolled But Not Randomized | Total
Number analyzed (Participants) | 3 | 4 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 2 | 8
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (8.1) | 52.3 (4.6) | 42.6 (10.4) | 52.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: To assess the safety and tolerability of bortezomib with mycophenolate mofetil assessed by the incidence of serious adverse events.
Time Frame: First dosing day to last study visit day: Mean duration 8 months.
Population: All subjects who received at least one dose.
Measure: Mean (Standard Deviation); unit: Number of Participants with Serious Adve
Arm/Group | Bortezomib Plus Mycophenolate Mofetil | Placebo Plus Mycophenolate Mofetil
Number analyzed (Participants) | 3 | 4
Number of Participants with Serious Adve | 0.33 (.58) | 0.25 (.50)

2. Secondary Outcome: Change of Skin Fibrosis Measured by the Rodnan Skin Score Between Baseline and 24 Weeks
Description: The Modified Rodnan Skin Score (mRSS) is a measure of skin thickness that sums individual scores of skin thickness (0 - No Thickening, 1 - Mild Thickening, 2 - Moderate Thickening, 3 - Severe Thickening) measured at 17 body sites to reach a total score (Range: 0 to 51, higher value representing thicker skin). The Score is used as a surrogate for disease activity and severity, and a worsening score over time is associated with worse outcomes.
Time Frame: 24 weeks
Population: All subjects who had comparable skin score data.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Bortezomib Plus Mycophenolate Mofetil | Placebo Plus Mycophenolate Mofetil
Number analyzed (Participants) | 3 | 3
Score on a Scale | -3.00 (2.65) | -0.33 (0.58)

3. Secondary Outcome: Change of Lung Function Measured by Forced Vital Capacity (FVC) Between Baseline and 24 Weeks
Description: Forced vital capacity, or FVC, is the amount in liters of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It measures the effect that lung disease has on a person's ability to inhale and exhale. Higher values are better, and decreases over time can indicate disease progression.
Time Frame: 24 weeks
Population: All subjects who had comparable forced vital capacity data.
Measure: Mean (Standard Deviation); unit: Percentage of change in FVC %predicted
Arm/Group | Bortezomib Plus Mycophenolate Mofetil | Placebo Plus Mycophenolate Mofetil
Number analyzed (Participants) | 3 | 3
Percentage of change in FVC %predicted | 0.51 (0.55) | -0.69 (1.02)

ADVERSE EVENTS:
Time Frame: First dosing day to last study visit day: Mean duration 8 months.
Description: Adverse event information collected by study team at each study visit.
Arm/Group | Bortezomib Plus Mycophenolate Mofetil | Placebo Plus Mycophenolate Mofetil
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib Plus Mycophenolate Mofetil (N=3) | Placebo Plus Mycophenolate Mofetil (N=4)
Herpes Zoster Infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Bilaterial Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib Plus Mycophenolate Mofetil (N=3) | Placebo Plus Mycophenolate Mofetil (N=4)
Ache on forehead and eyelids (General disorders) | 0 (0) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bach ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bruising at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burning sensation at injection site (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 1 (1)
Cold sweats (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough with increased mucus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 1 (1)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dry eyes (Eye disorders) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 3 (9) | 1 (2)
High cholesterol (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Left ankle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (14) | 0 (0)
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pain in right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pre-diabetes (Endocrine disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prolonged coughing episode (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Redness at injection site (Injury, poisoning and procedural complications) | 3 (6) | 0 (0)
Right side back muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Shaking (General disorders) | 1 (1) | 0 (0)
Skin peeling at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tingling at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Soreness at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tingling sensation on face (Nervous system disorders) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 1 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2)
Vomiting due to coughing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Warmth at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight loss of ~10 lbs (General disorders) | 1 (1) | 0 (0)
Worsened body aches (General disorders) | 0 (0) | 1 (1)
Worsened cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Worsened fatigue (General disorders) | 0 (0) | 1 (1)
Worsening diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT02370693/Prot_SAP_000.pdf